CLINICAL TRIAL: NCT04335344
Title: Evaluation of Plasma and Salivary suPAR in Periodontitis and CVD Patients
Brief Title: Role of suPAR in Periodontitis and CVD
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Collaborators: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Other Study IDs: 11-18-18
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Metabolic Disturbance; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Healthy patients
  Interventions: Other: Observation of suPAR plasma and salivary levels
- Periodontitis: Patients with periodontitis
  Interventions: Other: Observation of suPAR plasma and salivary levels
- Cardiovascular disease: Patients with cardiovascular disease
  Interventions: Other: Observation of suPAR plasma and salivary levels
- Periodontitis + cardiovascular disease: Patients with Periodontitis + cardiovascular disease
  Interventions: Other: Observation of suPAR plasma and salivary levels

INTERVENTIONS:
Other: Observation of suPAR plasma and salivary levels — Evaluation of suPAR plasma level and correlation of plasma suPAR levels with periodontal and cardiovascular disease

SUMMARY:
soluble urokinase-type plasminogen activator receptor (suPAR) plays a key role in endothelial function and may be a link for the known interaction of periodontitis and cardiovascular disease (CVD). The investigators compared the impact of gingival health, periodontitis (CP), CHD or of both diseases (CP+CHD) on saliva and serum suPAR levels.

DETAILED DESCRIPTION:
The aim of this study was to evaluate a possible association between both saliva and serum suPAR levels in patients with CP and with CVD and if the serum suPAR levels are mediated by serum CRP.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 15 teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL) ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects (n=33) and patients with periodontitis (n=35), CVD (n=34), and a combination of periodontitis + CVD (n=34) were enrolled in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2015-02-15 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 1-year
  evaluation of changes in clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matarese, Study Chair — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: 10 years at least
Access Criteria: Pubmed